CLINICAL TRIAL: NCT06558903
Title: Study of Predictive Biomarkers of Response to Carboplatin Etoposide Atezolizumab Combination in Patients With Small Cell Lung Cancer, Exploratory Study by HYPErionTM Tissue Mass Imaging
Brief Title: Searching for Predictive Biomarkers of Efficacy in Small Cell Lung Cancer Patients Treated With Chemotherapy-immunotherapy Combination Using Imaging Mass Cytometry (HYPE)
Acronym: HYPE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0110 - HYPE
Record Dates: First submitted 2024-08-09; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Biomarker; Immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Fixed tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective study is to identify predictive biomarkers of efficacy in tumor samples of small cell lung cancer patients treated with chemotherapy-immunotherapy combination using imaging mass cytometry. The main question it aims to answer is: is there any feature in the tumour microenvironment that can discriminate responders from non responders before treatment? Participants will provide consent for the collection of their clinical data and the study of their tumor samples

DETAILED DESCRIPTION:
Small cell lung cancer patients treated with first-line atezolizumab plus platinum-etoposide regimen with available formalin fixed paraffin embedded (FFPE) biopsies at baseline will be identified from Brest University Hospital medical records and their samples will be retrieved from Brest University Hospital Pathology Laboratory for imaging mass cytometry analyses.

Clinical data will be collected for each patient, including progression-free survival (defined as the time between treatment start and date of progression according to investigator, or death from any cause) and overall survival (defined as the time between treatment start and date of death from any cause).

For imaging mass cytometry analyses, a panel of 39 metal-tagged antibodies will be used to characterize the cell composition of lung tumors at baseline (inflammatory, tumor and stromal cells).

Statistical analyses will be performed to correlate the composition of the tumor microenvironment at baseline and the survival data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with extensive or metastatic small cell lung cancer
* Patients who started a first line treatment with atezolizumab plus carboplatin and etoposide in routine practice before February 2021
* Patients with available tumor sample before treatment start
* No objection from living patients

Exclusion Criteria:

* Patients who started first line treatment with atezolizumab plus carboplatin and etoposide in routine practice after February 2021
* Patients having received immunotherapy in a clinical trial
* Patients with auto-immune disorder
* Patients under legal protection (guardianship, curatorship)
* Patients refusing to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who started a first line treatment with atezolizumab plus carboplatin and etoposide at Brest University Hospital before February 2021 with available tumor sample before treatment start
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive biomarkers of anti-PD-L1 efficacy in the tumor of small cell lung cancer patients | 3 year
  Features in the tumour microenvironment that can discriminate patients responding to anti-PD-L1 from non responders

SECONDARY OUTCOMES:
Progression-free survival | 3 year
  Time between treatment start and date of progression according to investigator, or death from any cause
Overall survival | 3 year
  Time between treatment start and date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Geier, MD, Study Director — Department of Medical Oncology, Brest University Hospital; Pierre Le Noac'h, MD, Principal Investigator — Department of Medical Oncology, Brest University Hospital
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending five years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. requestors will be required to sign and complete a data access agreement